CLINICAL TRIAL: NCT02829736
Title: Pain and Reasons for Hospitalization in Patients Treated Without Post-operative Chest Tube After Thoracoscopic Wedge Resection - A Randomized Controlled Study
Brief Title: ThOracoscopic Wedge Resection Treated With Chest Tube Removal Intraoperatively
Acronym: TOTTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bo Laksáfoss Holbek, Medical doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-16028354
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Pain; Decreased Lung Function; Delayed Discharge
Keywords: lung neoplasm; lung metastasis; enhanced recovery after surgery; fast-track surgery; intraoperative chest tube removal; pain; lung function; reasons for admission
MeSH Terms: conditions — Pain; Respiratory Insufficiency; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Randomization occurs after ended surgery, thus masking allocation to the personnel and participant. After Randomization, there is no masking.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chest tube group (Active Comparator): Participants undergoing video-assisted thoracoscopic wedge resection with a positive intraoperative sealing test are treated with a standard post-operative chest tube.
  Interventions: Procedure: Intraoperative sealing test; Procedure: Standard post-operative chest tube
- No chest tube group (Experimental): Participants undergoing video-assisted thoracoscopic wedge resection with a positive intraoperative sealing test are treated with intraoperative chest tube removal.
  Interventions: Procedure: Intraoperative sealing test; Procedure: Intraoperative chest tube removal

INTERVENTIONS:
Procedure: Intraoperative sealing test — A standard 28 Fr chest tube is inserted through the anterior port hole and all port holes are closed. With the tip of the chest tube below water, the pleura is emptied from air during continuous ventilation of the lungs. An air leak after 5 minutes of ventilation indicates a negative sealing test, whereas a cessation of air leak within 5 minutes indicates a positive sealing test.
Procedure: Standard post-operative chest tube — A regular chest tube is left in the pleura.
  Arms: Chest tube group
Procedure: Intraoperative chest tube removal — Chest tube is removed intraoperatively.
  Arms: No chest tube group

SUMMARY:
Chest tubes are used routinely although preliminary studies demonstrate the feasibility and safety of intraoperative chest drain removal. Previous studies are however either retrospective or mainly concerning benign disease.

Hypothesis: Participants treated without post-operative chest tube after thoracoscopic wedge resection have less pain, better pulmonary function and similar complication profile than participants treated with standard post-operative chest tube, and could possibly be discharged earlier.

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracoscopic wedge resection
* Speaks and understands Danish
* FEV1 >= 60% of expected

Exclusion Criteria:

* Increased risk of air leak evaluated by surgeon (large adhesions, bullae, emphysema, deep resection, etc.)
* Increased risk of bleeding evaluated by surgeon (high INR, anticoagulation not paused, large bleeding, etc.)
* Air leak on intraoperative sealing test
* Patients previously included in study
* Planned intraoperative frozen section with possible lobectomy
* Previously included in current study
* Planned frozen section diagnostics
* Previous ipsilateral anatomic lung resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Pain | Through post-operative admission, an average of 1 day.
  Average pain expressed as area under the curve from a numeric rank score at 1, 3, 6 and 9 hours after surgery as well as daily at 8 am and 8 pm from post-operative day 1 until discharge.

SECONDARY OUTCOMES:
Reasons for post-operative admission | Through post-operative admission, an average of 1 day.
  Daily evaluation of reasons for admission.
Lung function | Up to post-operative day 1.
  FEV1 measured preoperatively and on post-operative day 1 at 8 am.
Reinsertion of chest tubes | Up to post-operative day 30.
  Frequency of chest tube reinsertion.
Pneumothorax | Up to post-operative day 1.
  Size and frequency of pneumothorax on x-ray after removal of chest tube
Complications | Up to post-operative day 30.
  Surgical complications including mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik J. Hansen, MD, Study Director — Rigshospitalet, Denmark; René H. Petersen, MD, Study Director — Rigshospitalet, Denmark; Henrik Kehlet, DMSc, Study Director — Rigshospitalet, Denmark; Bo L. Holbek, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No